CLINICAL TRIAL: NCT04665908
Title: PT-led Triage in Secondary Care Settings for Patients With Hip or/and Knee Osteoarthritis
Brief Title: PT-led Triage for Patients With Hip o Knee Osteoarthritis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Maziar Mohaddes Ardebili, MD Doctor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Triage and hip/knee OA
Record Dates: First submitted 2020-12-07; First posted 2020-12-14 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Knee Osteoarthritis; Hip Osteoarthritis
Keywords: PT-led triage; Osteoarthritis; Knee; Hip
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip; Osteoarthritis

STUDY DESIGN:
Masking Description: Due to the design of the study, it is not possible to blind either caregivers or participants regarding group distribution
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PT-led triage (Other): Patients are assessed by PT
  Interventions: Other: Assessment by PT/Orth surgeon
- Standard care (Other): The patiens are assessed by a orthopedic surgeon
  Interventions: Other: Assessment by PT/Orth surgeon

INTERVENTIONS:
Other: Assessment by PT/Orth surgeon — Assessment by orthopaedic surgeon or a PT

SUMMARY:
The aim of this project is to compare PT-led triage in secondary care setting for patients with hip or/and knee osteoarthritis (OA) with standard care (i.e. assessment of orthopedic surgeon). Comparison between cost-effectiveness, selection accuracy, patients perceived quality of care, quality of life and physical function will be made.

A further aim is to explore patients expectations and experiences of PT-led triage in a secondary care setting.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a common musculoskeletal disorder and the number of people in need of surgical treatment for hip and knee OA is increasing. The waiting time for consultation with an orthopedic surgeon (OS) is long and the majority of the patient referred for assessment are not appropriate for surgical intervention. To reduce the number of patients seen by an OS and thereby shorten the waiting time, Sahlgrenska University Hospital started a Physiotherapist-led (PT-led) triage project in 2017. With PT-led triage the patients are assessed by a physiotherapist to establish the most appropriate care management; if the patient is appropriate for surgery, should be referred for continued rehabilitation, or referred back to the referring physician. To our knowledge this model of care with PT-led triage in secondary care setting have not been scientifically evaluated in Sweden.

The aim of this project is to compare PT-led triage in a secondary care setting with standard care (i.e. assessment of OS for patients with knee or /and hip OA). A further aim is to determine if a digital triage tool can accurately predict when a primary knee or hip referral is deemed for nonsurgical versus surgical intervention by the surgeon following the first consultation.

Patients referred from primary care to Sahlgrenska University hospital with primary hip and/or knee OA will be included and randomized to consultation with either PT (triage) or OS (standard practice). Data about patient reported health-related quality of life, pain, function, and patients' perception of quality of care will be collected using questionnaires at baseline, 3 and 12 months after the consultation.

Data about waiting time for consultation, proportion of patients appropriate for surgery, further investigations, and data to be able to perform cost analysis will be collected from patients´ journals, the patient administration systems, both locally and via the region Västra Götaland´s database (VEGA).

A qualitative approach will be used to further investigate patients expectations and experience of a PT-led trige.

ELIGIBILITY:
Inclusion Criteria:

* Referred to Sahlgrenska University hospital
* Primary osteoarthritis in the hip or knee
* Understanding and speaking Swedish

Exclusion Criteria:

* Prior assessment by and referral from an orthopedic surgeon for the current problem
* Secondary osteoarthritis (posttraumatic osteoarthritis, femoral head necrosis), when stated on the referral
* Referred to a specific surgeon

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 675 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Short form of the Quality from Patients Perspective (QPP) | Baseline
  A Measure of patients' perception of quality of care regarding four dimensions: caregivers' medical-technical competence; care organizations' physical-technical conditions; degree of identity-orientation in the caregivers' attitudes and actions; and the care organizations' socio-cultural atmosphere

SECONDARY OUTCOMES:
Heath-related quality of life - EuroQol (EQ5-D) | Baseline, 3 and 12 months
  Measure of health-related quality of life and consists of 5 items. General health is measured using a VAS scale (0 to 100) with 100 being the best possible health state
Pain Disability index (PDI | Baseline, 3 and 12 months
  A questionnaire where respondents are asked to rate disability on a numeric rating scale ranging from 0 (no disability) to 10 (maximum disability) in seven areas; family and home responsibilities, recreation, social activity, occupation, sexual behavior, self-care, and life-support activity.
Forgotten Joint Score (FJS) | Basline, 3 and 12 months
  A questionnaire that was developed to find subtle differences between patients who grade their hip / knee as "very good" and "excellent". The score is graded from 0 to 100, where a high score is better
Oxford Hip/Knee Score (OHS/OHK | Basline, 3 and 12 months
  A questionnaire consisting of 12 questions that concern areas such as pain and disabilities the patient has experienced during the past four weeks.

OTHER OUTCOMES:
Patients expectations and experiences of PT-led triage | Interviews sep 2024-nov 2024
  Qualitative semistructured one to one interviews

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg, Västra Götaland County
  - Sahlgrenska University hospital, Gothenburg

REFERENCES:
- [Derived] Gustavsson L, Mohaddes M, Samsson K, Beischer S. No major difference in perceived quality of care in patients with hip or knee osteoarthritis assessed in a physical therapy-led triage compared with standard care: a randomized controlled trial. BMC Musculoskelet Disord. 2023 Jun 29;24(1):530. doi: 10.1186/s12891-023-06659-5. PMID 37386368